CLINICAL TRIAL: NCT02558517
Title: Evaluation of the Discontinuation of Maintenance Corticosteroid Treatment (Prednisone 5 Milligram Per Day) in Quiescent Systemic Lupus
Brief Title: Evaluation of the Discontinuation of Maintenance Corticosteroid Treatment in Quiescent Systemic Lupus
Acronym: CORTICOLUP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Dr Cohen Aubart, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: medint002
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Corticosteroids; Chronic disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone maintenance (No Intervention): Patients will be kept under Prednisone 5 milligrams/day. Other treatments will be maintained (in particular HYDROXYCHLOROQUINE, METHOTEXATE etc..)
- Prednisone discontinuation (Experimental): Prednisone will be stopped and remplaced by HYDROCORTISONE for one month (20 mg/day). Other treatments will be maintained (in particular HYDROXYCHLOROQUINE, METHOTEXATE etc..)
  Interventions: Drug: prednisone discontinuation

INTERVENTIONS:
Drug: prednisone discontinuation — randomization
  Other Names: prednisone maintenance
  Arms: Prednisone discontinuation

SUMMARY:
Systemic Lupus (SLE) is a chronic disease for which long term treatments are warranted. The aim of this study was to study the possibility of corticosteroids interruption in patients with quiescent SLE treated since at least one year with 5 milligrams of predonisone per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SLE according to the ACR revised criteria.
* Quiescent disease without flare since at least one year (SELENA SLEDAI < or equal to 4, BILAG C, D or E, PGA 0) _ Treatment with 5 milligrams/day of prednisone since at least 1 year

Exclusion Criteria:

* failure to sign the informed consent or unable to consent
* Patient participating to another clinical trial
* Pregnancy or plan to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of mild or moderate flares of SLE defined by the SLE FLARE Index | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zahir AMOURA, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière, Service de médecine Interne 2, Institut e3m, Paris, France

REFERENCES:
- [Derived] Mathian A, Pha M, Haroche J, Cohen-Aubart F, Hie M, Pineton de Chambrun M, Boutin THD, Miyara M, Gorochov G, Yssel H, Cherin P, Devilliers H, Amoura Z. Withdrawal of low-dose prednisone in SLE patients with a clinically quiescent disease for more than 1 year: a randomised clinical trial. Ann Rheum Dis. 2020 Mar;79(3):339-346. doi: 10.1136/annrheumdis-2019-216303. Epub 2019 Dec 18. PMID 31852672